CLINICAL TRIAL: NCT05642533
Title: Obesity and Cardiovascular Diseases, Cross-sectional Study in Saudi Arabia
Acronym: OCCURS
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-7510; U1111-1279-3716 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Obesity and Cardiovascular Risk
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Without a history of Type 2 diabetes: Adults with obesity
  Interventions: Other: No treatment given
- With a history of Type 2 diabetes: Adults with obesity
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
The purpose of this research study is to collect information on participants body weight, blood sugar levels, heart related diseases and lifestyle. The collected information will help estimate the prevalence of participants disease.

This study will take about 6 months. However, participants involvement in the study will not extend beyond their routine visit and will thus require a maximum of 1 day.

If participants choose to take part, they will be asked to give information about their health in routine clinical visit. Participants will be asked to complete a questionnaire about their lifestyle. Participants will complete this questionnaire during their normally scheduled visit with their doctor. Participants will continue their normal way of life and will not get any medication other than those prescribed to them by their doctor.

Participants will have no direct benefit from participation in this study and there are no risks involved.

Participants decide voluntarily whether they want to participate in this study or not. Participants' decision will not affect their medical care and they do not have to justify their decision.

Participants are free to leave the study at any time and without giving reasons. This does not affect their current or future treatment. The data collected up to that point are still being evaluated.

There is no additional cost to participants for being in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed consent obtained before any study related activities (study related activities are any procedure-related to recording of data according to the protocol).
2. Diagnosed with obesity (BMI higher than or equal to 30 for all ethnic groups except Asian; BMI higher than or equal to 27.5 for patients of Asian ethnicity).
3. Diagnosed with T2D for patients in Cohort 2.
4. Male or female, aged between 18 and 75 years at the time of signing informed consent

Exclusion Criteria:

1. Participation in an interventional clinical trial during the study period.
2. Diagnosed with T2D for patients in Cohort 1.
3. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adults with obesity, either without a history of T2D (Cohort 1) or with a history of T2D (Cohort 2).
Sampling Method: Non-Probability Sample
Enrollment: 1061 (Actual)
Dates: Start 2022-12-31 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Proportion of people with obesity without a history of Type 2 diabetes (T2D) who have Cardiovascular disease (CVD)s (pre-existing or newlydiagnosed) | At time of patient enrollment/cross-sectional routine visit (DAY 1)
  Percentage (and 95% confidence interval [CI])

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com